CLINICAL TRIAL: NCT02668991
Title: A Study to Assess the Janssen Autism Knowledge Engine in Children and Adults With Autism Spectrum Disorder and in a Normally Developing Cohort
Brief Title: Study to Assess the Janssen Autism Knowledge Engine in Participants With Autism Spectrum Disorder and in a Normally Developing Cohort
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR106701; MENTIS-ASD002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Janssen Autism Knowledge Engine; Autism Behavior Inventory
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: It will consist of planned 100 children and adults with Autism Spectrum Disorder (ASD) aged 6 years and older with no requirements regarding concurrent therapies or treatments.
- Cohort 2: It will consist of planned 50 children and adults aged 6 and older who, as part of their standard care, happen to be beginning a behavioral intervention within 2 weeks after the baseline visit of the study. This intervention can be an applied behavior analysis (ABA) program or similar or a social skills program or a school-based autism program and must be intended to last at least throughout the duration of the study.
- Cohort 3: It will consist of planned 30 normally developing children and adults. These participants will only have a single visit wherein they will undergo a single session with the task battery and biosensors. There should be 5 participants aged 6-9 years, 5 aged 10-12 years, 5 aged 13-17 years, and 5 aged 18 years and older. This cohort should approximate the male:female ratio in Cohorts 1 & 2, with approximately 1 female for every 5 males.

SUMMARY:
The purpose of this study is to evaluate the utility of and to clinically validate the Autism Behavior Inventory (ABI) in measuring clinical symptoms of Autism Spectrum Disorder (ASD) compared with other gold standard measures.

DETAILED DESCRIPTION:
This is an observational study (in which participants identified as belonging to study groups are assessed for biomedical or health outcomes) to evaluate the utility of Janssen Autism Knowledge Engine (JAKE) in measuring clinical symptoms of ASD in children and adults with ASD. The study will consist of 3 cohorts of participants. For Cohort 1 and 2, there will be 14-day Screening phase and 8-week (Cohort 1) or 10 week (Cohort 2) data collection phase extending from Day 0 (Baseline) to Day 56 or Day 70, respectively. For Cohort 3, the study will consist of a screening visit and a single testing visit, which may be combined. Primarily, the usability of JAKE as a system to monitor clinical outcomes in ASD will be assessed. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 and 2:

* Participants must be males or females aged 6 years and older with at least one female for every five male participants
* Diagnosis of ASD made or confirmed using the Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2)
* Participants can receive behavioral and/or pharmacologic treatments for ASD and comorbid disorders during the course of the study, or not (Cohort 1)
* In cohort 2, as part of their standard care participants must be about to begin a behavioral intervention within 2 weeks after the Baseline visit
* Parents or legally authorized representatives must speak and understand English

Cohort 3:

* Participants must be males or females aged 6 years and older with at least one female for every five male participants.
* Parents or legally authorized representatives must speak and understand English
* In the opinion of the investigator, subject and parents must be capable of completing all procedures and tasks of the study
* Each participant or their legally authorized representative must sign an informed consent form (ICF)
* A score in the normal range on the Social Communication Questionnaire (SCQ) and must not have any Diagnostic and Statistical Manual of Mental Disorders

Exclusion Criteria:

Cohort 1 and 2:

* Measured composite score on the Kaufmann Brief Intelligence Test-2 (KBIT-2) of less than 60
* History of, or current significant medical illness that the Investigator considers should exclude the participant
* Psychological and/or emotional problems which would render the informed consent invalid or limit the ability of the subject to comply with the study requirements
* Any condition that in the opinion of the investigator would compromise the study, or the wellbeing of the subject; for example, visual problems that would impede eye-tracking or viewing the stimuli or hearing problems that would impede hearing auditory stimuli
* Participant is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator

Cohort 3:

* History of or current significant medical illness that the Investigator considers should exclude the participant
* Psychological and/or emotional problems which would render the informed consent invalid or limit the ability of the participant to comply with the study requirements
* Any condition that in the opinion of the investigator would compromise the study, or the wellbeing of the subject; for example, visual problems that would impede eye-tracking or viewing the stimuli or hearing problems that would impede hearing auditory stimuli
* Participant is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator
* Participant should not take any sedating medications on the day of the test battery and should not consume caffeine within 2 hours prior to the battery

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and Adult participants with history of Autism Spectrum Disorder (ASD) will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Utility of Autism Behavior Inventory(ABI) in Measuring Clinical Symptoms of Autism Spectrum Disorder (ASD) | up to Week 10
  The ABI is a series of 73 questions related to the core and associated symptoms of ASD. Questions are answered on two 4-point scales, consisting of ratings of frequency and intensity, frequency and context, or quality and context.

SECONDARY OUTCOMES:
Usability of the Janssen Autism Knowledge Engine (JAKE) in Measuring Clinical Symptoms of ASD | up to Week 10
  The JAKE personal healthcare record (pHR) encompasses various modules for use by clinicians, caregivers, participants and the sponsor. The JAKE is accessible both through a web interface for computers and applications for mobile devices. The modules are Medical/Developmental History, Autism Behavior Inventory (ABI), Journal/ASD events, Treatment Tracker, Dashboard, HealthVault, Research Data Warehouse and Workbench. Results of several parent and clinician questionnaires will be compared with the findings of the mentis ABI and biosensors. An exit survey will assess overall usability of the system.
Correlation Between Key Biosensors and Autism Spectrum Disorder (ASD) Symptoms | up to Week 10
  The utility of the biosensors will be determined by measuring the associations between the biosensors and the ASD symptoms (response to tasks and stimuli in lab, the ABI, standard scales, and the event tracker).
Correlation Between Genomic Characteristics and Autism Phenotypes | up to Week 10
  Genomic analysis will be done by analyzing DNA samples related to the JAKE System or autism spectrum disorder.
Usability of the JAKE System to detect changes in response to standard | up to Week 10
  Change is symptoms in response to coincident courses of treatment with standard behavioral therapy as measured with the JAKE system.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to Week 10
Normative data on the JAKE Biosensor Array (Continuous and Periodic) | up to Week 10
  Normative data on the JAKE biosensor array (Continuous and Periodic) will be collected. Comparisons between Cohort 3 and Cohorts 1 and 2 will be made to examine differences between normally developing and ASD participants.
Normative data on the JAKE Task Battery | up to Week 10
  Normative data on the JAKE task battery will be collected. Comparisons between Cohort 3 and Cohorts 1 and 2 will be made to examine differences between normally developing and ASD participants.
Ease of use of JAKE for use in Prospective Clinical Trials | up to Week 10
  The JAKE personal healthcare record (pHR) encompasses various modules for use by clinicians, caregivers, participants and the sponsor. The JAKE is accessible both through a web interface for computers and applications for mobile devices. The modules are Medical/Developmental History, ABI, Journal/ASD events, Treatment Tracker, Dashboard, Health Vault, Research Data Warehouse and Workbench.
Utility of JAKE for use in Prospective Clinical Trials | up to Week 10
  The JAKE personal healthcare record (pHR) encompasses various modules for use by clinicians, caregivers, participants and the sponsor. The JAKE is accessible both through a web interface for computers and applications for mobile devices. The modules are Medical/Developmental History, ABI, Journal/ASD events, Treatment Tracker, Dashboard, Health Vault, Research Data Warehouse and Workbench.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (9):
- United States (9):
  - Phoenix, Arizona
  - San Francisco, California
  - New Haven, Connecticut
  - Worcester, Massachusetts
  - Toms River, New Jersey
  - Orangeburg, New York
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Seattle, Washington

REFERENCES:
- [Derived] Kaliukhovich DA, Manyakov NV, Bangerter A, Pandina G. Context Modulates Attention to Faces in Dynamic Social Scenes in Children and Adults with Autism Spectrum Disorder. J Autism Dev Disord. 2022 Oct;52(10):4219-4232. doi: 10.1007/s10803-021-05279-z. Epub 2021 Oct 8. PMID 34623583
- [Derived] Kaliukhovich DA, Manyakov NV, Bangerter A, Ness S, Skalkin A, Goodwin MS, Dawson G, Hendren RL, Leventhal B, Hudac CM, Bradshaw J, Shic F, Pandina G. Social attention to activities in children and adults with autism spectrum disorder: effects of context and age. Mol Autism. 2020 Oct 19;11(1):79. doi: 10.1186/s13229-020-00388-5. PMID 33076994
- [Derived] Bangerter A, Manyakov NV, Lewin D, Boice M, Skalkin A, Jagannatha S, Chatterjee M, Dawson G, Goodwin MS, Hendren R, Leventhal B, Shic F, Ness S, Pandina G. Caregiver Daily Reporting of Symptoms in Autism Spectrum Disorder: Observational Study Using Web and Mobile Apps. JMIR Ment Health. 2019 Mar 26;6(3):e11365. doi: 10.2196/11365. PMID 30912762
- [Derived] Ness SL, Bangerter A, Manyakov NV, Lewin D, Boice M, Skalkin A, Jagannatha S, Chatterjee M, Dawson G, Goodwin MS, Hendren R, Leventhal B, Shic F, Frazier JA, Janvier Y, King BH, Miller JS, Smith CJ, Tobe RH, Pandina G. An Observational Study With the Janssen Autism Knowledge Engine (JAKE(R)) in Individuals With Autism Spectrum Disorder. Front Neurosci. 2019 Feb 27;13:111. doi: 10.3389/fnins.2019.00111. eCollection 2019. PMID 30872988